CLINICAL TRIAL: NCT02891980
Title: A Phase I Trial to Utilize Systems Biology Approaches to Examine the Safety, Immunogenicity, and 'Omics Response to MVA-BN(R)-Filo and Ad26.ZEBOV Vaccines in Healthy Volunteers
Brief Title: A Safety Trial to Test MVA-BN(R)-Filo and Ad26.ZEBOV Vaccines in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0094
Record Dates: First submitted 2016-09-01; First posted 2016-09-08 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2017-07-19

CONDITIONS: Ebola Disease; Marburg Disease
Keywords: Ad26.ZEBOV; Ebola; Immunogenicity; Marburg; MVA-BN-Filo; Omics; Zaire
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Marburg Virus Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 2 (Experimental): MVA-BN®-Filo Day 1, Ad26.ZEBOV Day 29 and MVA-BN®-Filo Day 366
  Interventions: Biological: Ad26 Zaire Ebola Vaccine; Biological: MVA Multi-Filo Ebola Vaccine
- Group 3 (Experimental): Ad26.ZEBOV Day 1, MVA-BN®-Filo Day 29 and MVA-BN®-Filo Day 366
  Interventions: Biological: Ad26 Zaire Ebola Vaccine; Biological: MVA Multi-Filo Ebola Vaccine
- Group 4 (Experimental): Ad26.ZEBOV Day 1, Ad26.ZEBOV Day 29
  Interventions: Biological: Ad26 Zaire Ebola Vaccine
- Group1 (Experimental): MVA-BN®-Filo Day 1 and MVA-BN®-Filo Day 29
  Interventions: Biological: MVA Multi-Filo Ebola Vaccine

INTERVENTIONS:
Biological: Ad26 Zaire Ebola Vaccine — A recombinant adenovirus vector comprising a polynucleotide encoding a filovirus antigenic protein, wherein the recombinant adenovirus vector comprises an adenovirus 26 capsid protein.
  Arms: Group 2; Group 3; Group 4
Biological: MVA Multi-Filo Ebola Vaccine — A multivalent MVA-BN Filovirus vaccine, designed to protect against Ebola Zaire, Ebola Sudan and Marburg virus.
  Arms: Group 2; Group 3; Group1

SUMMARY:
This is a Phase 1, double-blind, randomized trial to evaluate the safety and immunogenicity of two heterologous and two homologous prime-boost regimens using MVA-BN(R)-Filo and Ad26.ZEBOV administered in different sequences at Days 1 and 29 in healthy adult subjects aged 18 - 45 years. The study will evaluate the 'omics (transcriptomics, proteomics, lipidomics, metabolomics), antibodies for immunogenicity, CMI, ADCC, and plasmablast responses to MVA-BN(R)-Filo and Ad26.ZEBOV vaccines. The primary objectives of this study are: 1) To assess the safety and reactogenicity of each study group. 2) To assess responses to the study vaccination by study group after the first, second and third dose by transcriptomics. 3) To assess the peak antibody response to the study vaccination by study group to filovirus antigens.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized trial to evaluate the safety and immunogenicity of two heterologous and two homologous prime-boost regimens using MVA-BN(R)-Filo and Ad26.ZEBOV administered in different sequences at Days 1 and 29 in healthy adult subjects aged 18 - 45 years. The two heterologous prime-boost groups will also receive MVA-BN(R)-Filo at day 366. Sixty subjects will be randomized 1:1:1:1 to one of four study groups (15 per group). Subjects and study staff will be blinded to a subject's study vaccine assignment within study vaccination schedule (e.g., enrollment into Group 1 or 4 versus 2 or 3 will be known). The study will evaluate the 'omics (transcriptomics, proteomics, lipidomics, metabolomics), antibodies for immunogenicity, CMI, ADCC, and plasmablast responses to MVA-BN(R)-Filo and Ad26.ZEBOV vaccines. The primary objectives of this study are: 1) To assess the safety and reactogenicity of each study group. 2) To assess responses to the study vaccination by study group after the first, second and third dose by transcriptomics. 3) To assess the peak antibody response to the study vaccination by study group to filovirus antigens. Secondary objectives are: 1) To assess antigen-specific cell-mediated immune (CMI) responses to the study vaccination by study group. 2) To assess antibody-dependent cell-mediated cytotoxicity (ADCC) responses to the study vaccination by study group.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read and provide consent after completing the informed consent process.
2. Subject must be able to understand and comply with planned procedures.
3. Subject must be a man or woman aged > / = 18 to < / = 45 years.
4. Subject must have a body mass index (BMI) > / = 18.5 and < 35 kg/m^2.
5. Subject must be healthy on the basis of patient-reported medical history, physical examination, and the investigator's clinical judgment.
6. Subject must have acceptable laboratory parameters* within 28 days of enrollment:

   * Note 1: If the following acceptable screening laboratory parameters** are out of range, repeat of screening tests is permitted once, provided there is an alternative explanation for the out of range value. The alternative explanation for the out of range value should be documented in the subject's source documents. The acceptable value for repeated screening tests must be available within the 28 days screening period.

Acceptable laboratory parameters include the following:

* Hemoglobin: women: > / = 11.5 g/dL; men > / = 12.5 g/dL
* White blood cell (WBC) count: > 3.7 Thousand/uL but < 10.9 Thousand/uL
* Absolute neutrophil count > 1,500 cells/uL
* Platelets: > 139 but < 550 Thousand/uL
* Urinalysis (clean urine sample)*: protein and blood < 1+, glucose negative *Note: for women: in case of menstruation, urinalysis must be postponed, but a result should be available before Day 1.
* Alanine aminotransferase (ALT) < / = 1 x institutional upper limit of normal
* Serum creatinine < / = 1 x institutional upper limit of normal
* Troponin I < / = 1 x institutional upper limit of normal
* Fibrinogen > 140 mg/dL but < / = 500 mg/dL
* Prothrombin time (PT) < / = 1 x institutional upper limit of normal
* Activated partial thromboplastin time (PTT) < / = 1 x institutional upper limit of normal.
* Negative test for HIV.
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.

  * Note 2: Grade 1 abnormalities for laboratory tests other than those covered in this list are considered acceptable if not clinically significant. If a Grade 2 or Grade 3 abnormality for lab tests other than those covered in this list is identified, repeating the screening tests is permitted once provided there is an alternative explanation for the out-of-range value. The alternative explanation for the out of range value should be documented in the subject's source documents.

    7. Women of childbearing potential must have a negative serum pregnancy test during screening and a negative urine pregnancy test immediately prior to each study vaccine administration.

    8. Women of childbearing potential must have an acceptable method of contraception* from 28 days before the prime vaccination until at least 3 months after the last boost vaccination.

    *Acceptable methods of birth control include the following:

    a. Prescription oral contraceptives, contraceptive injections, intrauterine device (IUD), implants, vaginal ring, double-barrier method, contraceptive patch, male partner sterilization b. Abstinence (defined as refraining from heterosexual intercourse) c. If not heterosexually active at screening, must agree to practice adequate birth control measures if they become heterosexually active from the start of screening onwards until at least 3 months after the last boost vaccination.

    d. Women of non-childbearing potential, defined as postmenopausal (any age with amenorrhea for > / = 6 months and serum follicle-stimulating hormone [FSH] > 40 mIU/mL) or surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), are not required to use the required birth control methods.

    9. Female subject agrees to not donate eggs (ova, oocytes) for the purposes of assisted reproduction from the start of screening onwards until at least 3 months after the last boost vaccination.

    10. Male subject who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use an acceptable method* of birth control until at least 3 months after the last boost vaccination.

    *Acceptable methods of birth control include the following:
    1. A double-barrier method of birth control, such as condom and partner with occlusive cap (diaphragm, cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
    2. In case the female partner is using an adequate method of birth control (see Inclusion Criterion #8), a single barrier method of birth control for the male subject is acceptable.

       11. Male subject must also agree not to donate sperm for the purposes of assisted reproduction from the start of screening onwards until at least 3 months after the last boost vaccination.

       12. Subject must be available and willing to participate for the duration of the study visits and follow-up (up to 19 months from enrollment).

       13. Subject must provide identification. 14. Subject must have a means to be contacted. 15. Subjects must have consistent access to the internet to perform electronic data entry.

       Exclusion Criteria:
       1. Has been vaccinated with an Ebola vaccine.
       2. Has been diagnosed with Ebola disease, or exposed to Ebola including travel to West Africa* in 2014-2016.

          * Note: West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone. Subjects who anticipate traveling to epidemic Ebola areas before the end of the study will also be excluded from enrollment into the study.
       3. Known or suspected receipt of an adenovirus serotype 26 (Ad26)-based vaccine.
       4. Known or suspected receipt of any licensed or investigational small pox (vaccinia)-based vaccine* *Note: Includes any MVA-based candidate vaccine (Imvamune or Imvanex), Dryvax, or Acam2000. Military history should be reviewed with potential subjects for receipt of vaccinia-based vaccine. The presence of a typical vaccinia scar should be considered exclusionary.
       5. Positive serology for human immunodeficiency virus (HIV)
       6. Positive Hepatitis B surface antigen
       7. Positive antibody to Hepatitis C virus (HCV)
       8. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products*.

          *Note: This includes a known allergy to egg, egg products and aminoglycosides or any of the constituents of the study vaccines [e.g., polysorbate 80, ethylenediaminetetraacetic acid (EDTA), L-histidine, tris (hydroxymethyl)-amino methane (THAM)).
       9. Has an acute illness or temperature > / = 38.0 degrees Celsius within the 3 days prior to Day 1.* *Note: Potential subjects can be rescheduled due to acute illness within the 28 day window between screening and enrollment. If acute illness prevents administration of vaccine within the 28 day screening window, the potential subject can be enrolled once the acute illness resolves after repeating safety laboratories and if the subject is otherwise eligible. The ECG does not need to be repeated as it is not a safety laboratory and unlikely to change without clinical event in this age group of volunteers.
       10. Female subject is pregnant or breast-feeding, or planning to become pregnant while enrolled in the study or within 3 months after the last boost vaccination.
       11. A history of bleeding or clotting disorders.
       12. Any clinically significant acute or chronic medical condition* that, in the opinion of the investigator, would preclude participation.

           * E.g., history of seizure disorders, autoimmune disease, immunodeficiency, any spleen disease, active malignancy, active tuberculosis, asthma, or other systemic infections.
       13. History of malignancy other than squamous cell or basal cell skin cancer*, unless there has been surgical excision that is considered to have achieved cure.

           * Note: Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
       14. Prior organ and/or stem cell transplant.
       15. Major surgery (per the investigator's judgment) within the 4 weeks prior to study entry or planned major surgery through the course of the study.
       16. History of myocarditis, pericarditis, cardiomyopathy, transient ischemic attack or stroke, myocardial infarction, angina, coronary artery disease, congestive heart failure, or arrhythmia*.

           *Note: This includes any clinically significant arrhythmia requiring medication, treatment, or clinical follow-up.
       17. Electrocardiogram (ECG) with clinically significant findings,* or features that would interfere with the assessment of myocarditis/pericarditis.

           *Clinical significant findings include the following:

    a. Conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS > / = 120 ms, PR interval > / = 210 ms, any second- or third-degree atrioventricular block, or prolongation of the QT interval corrected according to Bazett's formula [QTcB] [> 450 ms]) b. Significant repolarization (ST-segment or T-wave) abnormality. c. Significant atrial or ventricular arrhythmia; frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, 2 premature ventricular contractions in a row).

    d. ST-elevation consistent with ischemia or evidence of past or evolving myocardial infarction.

    18. History of diabetes mellitus type 1 or type 2*, including cases controlled with diet alone.
    * Note: A history of isolated gestational diabetes is not an exclusion criterion. 19. Thyroidectomy or thyroid disease requiring medication during the last 12 months.

      20. Uncontrolled hypertension, defined as systolic blood pressure > / = 140 mmHg or diastolic blood pressure > / = 90 mmHg.*
    * Note: Vital signs must be normal by protocol toxicity grading scale or determined to be normal-variant by investigator. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate may be re-measured. Repeated vital signs may be used to determine eligibility.

      21. Received a licensed live vaccine within 30 days prior to enrollment in this study, or plans to receive a licensed live vaccine within 30 days before or after each study vaccine.

      22. Received a licensed inactivated vaccine within 14 days prior to enrollment in this study, or plans to receive a licensed inactivated vaccine within 14 days before or after each study vaccine.

      23. Use of experimental therapeutic agents within 3 months from the start of screening.

      24. Current or planned participation in another clinical study during the study period.*
    * Note: Participation in an observational clinical study is allowed. 25. Receipt of blood products or immunoglobulin in the past 3 months. 26. Donation of a unit of blood within 8 weeks before Day 1 or plans to donate blood during participation in the study (from the start of screening onwards).

      27. Major psychiatric illness during the past 12 months that in the opinion of the investigator would preclude participation.

      28. Current or past abuse of recreational or narcotic drugs.*
    * Note: Urine will be tested only at screening to check for use of amphetamines, benzodiazepines, cocaine, and opioids.

      29. Current or past alcohol use judged by the investigator to potentially interfere with subject study adherence.

      30. History of chronic urticaria (recurrent hives). 31. Chronic or recurrent use of medications which modify host immune response (e.g., cancer chemotherapeutic agents, parenteral corticosteroids).*
    * Note: This is defined as greater than 2 weeks duration within three months prior to vaccination or current use of immunosuppressive medication:

      a. Permissible use during study include: corticosteroid nasal sprays for allergic rhinitis and low dose inhaled corticosteroids defined as < 800 mcg/day of beclomethasone dipropionate CFC or equivalent.

      b. Topical steroid for mild uncomplicated dermatitis such as poison ivy or contact dermatitis should be completed before study.

      c. Oral/parenteral corticosteroids given for non-chronic conditions not expected to recur are permissible if the length of therapy was < / = 14 days with completion at least 30 days prior to enrollment.

      32. Subject who cannot communicate reliably with the investigator. 33. Subject who, in the opinion of the investigator, is unlikely to adhere to the requirements of the study.

      34. Any condition that, in the opinion of the investigator, might interfere with assessing the study objectives.

      35. Personnel involved in the study*.
    * Note: This includes the Principal Investigator (PI), sub-Investigators listed in Form FDA 1572 or Investigator of Record Form, all staff who are paid entirely or partially by/through the OCRR contract for the trial, and staff who are supervised by the PI or sub-Investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Determine the differential expression from baseline in mRNA after each study vaccination by study group | Screening and Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 for Groups 1 and 4; additionally Days 366, 367, 369, 373, 380, 394, and 546 for Groups 2 and 3.
Determine the number of subjects with a vaccine-related serious adverse event (SAE) from the time of first study vaccination by study group through the duration of the study | Day 1 through Day 366 in Groups 1 and 4; Day 1 through Day 546 in Groups 2 and 3
Determine the number of subjects with a vaccine-related unsolicited adverse event (AE) from the time of each study vaccination by study group | Day 1 through Day 29
Determine the number of subjects with solicited local and systemic reactogenicity events from the time of study vaccination by study group. | Day 1 through Day 8
Determine the peak antibody response against filovirus glycoproteins (GPs) for each study group | Days 1, 15, 29, 36, 43, 57, 209, and 366 for Groups 1 and 4; additionally Days 369, 373, 380, 394, 546 for Groups 2 and 3.

SECONDARY OUTCOMES:
Determine the change in CMI response from baseline against filovirus antigen using peptide pools and measurement by intracellular cytokine staining (ICS) in each of the study groups | Days 1, 15, 29, 36, 43, 57, 209, and 366 in Groups 1 and 4; additionally Days 369, 373, 380, 394, and 546 in Groups 2 and 3.
Determine the change in the ADCC from baseline in each of the study groups | Days 1, 15, 29, 36, 43, 57, 209, and 366 for Groups 1 and 4; additionally Days 373, 380, 394, and 546 for Groups 2 and 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Rostad CA, Yildirim I, Kao C, Yi J, Kamidani S, Peters E, Stephens K, Gibson T, Hsiao HM, Singh K, Spearman P, McCracken C, Agbakoba V, Tomashek KM, Goll JB, Gelber CE, Johnson RA, Lee S, Maner-Smith K, Bosinger S, Ortlund EA, Chen X, Anderson LJ, Wrammert J, Suthar M, Rouphael N, Anderson EJ. A Phase 1 randomized trial of homologous and heterologous filovirus vaccines with a late booster dose. NPJ Vaccines. 2024 Dec 23;9(1):255. doi: 10.1038/s41541-024-01042-4. PMID 39715748